CLINICAL TRIAL: NCT01721733
Title: A Phase 2B Randomized, Placebo Controlled, Double Blind Clinical Trial of EPI-743 in Children With Leigh Syndrome
Brief Title: Safety and Efficacy Study of EPI-743 in Children With Leigh Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: Axio Research. LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPI743-12-002
Record Dates: First submitted 2012-11-01; First posted 2012-11-06 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Leigh Syndrome
Keywords: EPI743; Leigh syndrome; respiratory chain disease; mitochondrial disorders
MeSH Terms: conditions — Leigh Disease; Mitochondrial Diseases | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Each patient will receive a volume of placebo based on weight
  Interventions: Drug: Placebo
- EPI-743 15 mg/kg (Active Comparator): Each subjects dose will be based on their weight. 15 mg/kg with a maximum dose of 200 mg per dose, t.i.d., will be administered in this treatment arm.
  Interventions: Drug: EPI-743 15 mg/kg
- EPI-743 5 mg/kg (Active Comparator): Each subjects dose will be based on their weight. 5 mg/kg with a maximum dose of 100 mg per dose, t.i.d., will be administered in this treatment arm.
  Interventions: Drug: EPI-743 5 mg/kg

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: EPI-743 15 mg/kg
  Arms: EPI-743 15 mg/kg
Drug: EPI-743 5 mg/kg
  Arms: EPI-743 5 mg/kg

SUMMARY:
The purpose of this study is to evaluate the effects of EPI-743 in children with Leigh syndrome on disease severity, neuromuscular function, respiratory function, disease morbidity and mortality and disease associated biomarkers.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects of EPI-743 in patient with Leigh syndrome on disease severity, neuromuscular function, respiratory function, disease morbidity and mortality and biomarkers associated with the disease.

This study is a six month prospective randomized double-blind, placebo-controlled trial with a six month extension phase of two dose levels of EPI743. The planned enrollment is for approximately 30 children with genetically confirmed Leigh syndrome. After 6 months of treatment, those children that were randomized to the placebo treatment arm will be re-randomized to one of the 2 active treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and MRI diagnosis of Leigh syndrome
* Moderate disease severity based on NPMDS score
* Age under 18 years
* Documented evidence of disease progression within 12 month of enrollment
* Availability of MRI that confirms necrotizing encephalopathy
* Patient or guardian able to consent and comply with protocol requirements
* Abstention from Coenzyme Q10, Vitamins C & E, lipoic acid and Idebenone

Exclusion Criteria:

* Allergy to EPI-743, Vitamin E or sesame oil
* History of bleeding abnormalities or abnormal PT/PTT
* Diagnosis of concurrent inborn error of metabolism
* Previous tracheostomy
* Ventilator dependent or use of noninvasive ventilatory support w/in 1 month of enrollment
* LFTs greater than 2 times ULN
* Renal insufficiency
* End stage cardiac failure
* Fat malabsorption syndrome
* Use of anticoagulant medications
* Abstention from Botox for 6 months prior to enrollment and for duration of study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-05-31 (Actual)

PRIMARY OUTCOMES:
Newcastle Pediatric Mitochondrial Disease Scale (NPMDS) Sections 1-3 | 6 months
  Change from baseline to six months will be compared between subjects in active treatment group and placebo group

SECONDARY OUTCOMES:
Neuromuscular function | 6 months
  Gross Motor Function Measure; Barry Albright Dystonia Scale
Respiratory function | 6 months
  Need for tracheostomy
Disease morbidity | 6 months
  Total number of hospitalizations
Glutathione cycle biomarkers | 6 months
  Blood levels of glutathione will be compared between placebo and treatment group
Number of dose limiting serious adverse events | 6 months
Mortality | 6 months
  Number of deaths

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - Akron Children's Hospital, Akron, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Edison Pharmaceuticals Web Site — http://www.edisonpharma.com